CLINICAL TRIAL: NCT05336266
Title: IIT2021-16-Hendifar-KetoROCX: A Feasibility Study of Ketorolac Treatment for Cachexia in Patients With Advanced Pancreatic Ductal Adenocarcinoma
Brief Title: A Feasibility Study of Ketorolac Treatment for Cachexia in Patients With Advanced Pancreatic Ductal Adenocarcinoma
Acronym: KetoROCX
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Andrew Hendifar, MD (Other)
Collaborators: Yinuoke Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Andrew Hendifar, MD, Assistant Professor, Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2021-16-HENDIFAR-KETOROCX
Record Dates: First submitted 2022-03-11; First posted 2022-04-20 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Pancreas Cancer; Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer
Keywords: ketorolac
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketorolac (open label) (Experimental): Pancreatic patients receiving Ketorolac four times a day for up to five days
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Trial treatment of ketorolac 10mg orally four times a day for 5 consecutive days

SUMMARY:
The purpose of this study is to see if taking ketorolac, a nonsteroidal anti-inflammatory drug (NSAID), is reasonable, safe and can stabilize or increase weight along with quality of life in pancreatic cancer patients.

DETAILED DESCRIPTION:
The main things that will happen in this study are: patients will be administered ketorolac for 5 days, blood draws, completion of questionnaires, monitoring physical activity and sleep by wearing a study-provided FitBit along with weight using a study-provided smart scale.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of advanced and refractory pancreatic ductal adenocarcinoma (PDAC) referred to Cedars-Sinai Medical Center (CSMC).
2. Cachexia defined as ≥5% weight loss in the presence of chronic illness, within any 6-month period prior to screening or as documented by the medical physician based on standard diagnosis of cachexia.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 or Karnofsky performance status >50%.
4. Patient must have adequate renal function per below lab values:

   * Creatinine OR measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine or CrCl) ≤1.5 × upper limit of normal OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN.
5. Patient must have access to WiFi for the Smart Scale.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements in the opinion of the investigator.
2. Pregnancy, breastfeeding, or of childbearing potential and not willing to use adequate methods of contraception during the study.
3. Has any known allergies or hypersensitivity to the study drug or allergic reactions to surgical steel or elastomer/rubber.
4. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
5. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
6. Concurrent use of any other NSAIDs while on study.
7. Active peptic ulcer disease, recent gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding.
8. Have suspected or confirmed cerebrovascular bleeding, tendency to bleed or bruise easily, incomplete hemostasis (how you body stops bleeding), and at high risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility determined by the number of patients that take the prescribed dose of ketorolac (4 times daily) for 5 consecutive days. | 6 days
  Defined as 75% or more of patients taking the study medication as prescribed for 5 days in a 6-day period: compliance diary.

SECONDARY OUTCOMES:
To describe the adverse events associated with ketorolac when administered. | 14 days
  -Safety is defined as stable or decreased number of adverse events (AEs) compared to published trials for the same chemotherapy.
Mean change in weight from baseline through the End-of-Study visit | 14 days
  -Body weight stability is defined as weight change < 0.1kg/baseline Body Mass Index-unit from Baseline (start of 1 week lead-in prior to Day 1) to Day 6. Weight will be measured using the Aria Smart Scale. Changes in weight from Day 6 to Day 14 and from Day 1 to Day 14 will also be evaluated long term.
Mean change in body fat from baseline through the End-of-Study visit | 14 days
  -Body fat percentage will be measured using the Aria smart scale and compared from Baseline (start of 1 week lead-in prior to Day 1) to Day 6. Changes in body fat percentage from Day 6 to Day 14 and from Day 1 to Day 14 will also be evaluated long term. An increase in body fat percentage will be regarded as a positive outcome.
Evaluate change in quality of life including pain assessment from baseline through the End-of-Study visit | 14 days
  * Mean change in reported pain, sleep disturbance, and mood (anxiety/depression) using the NIH PROMIS-29 profile v2.1.
  * The PROMIS-29 profile v2.1 questionnaire consists of 29 questions that ask the subject to rate : 1) how easy it is to perform routine tasks, 2) how mood impacts daily living, 3) quality of sleep, 4) feelings of fatigue, and 5) pain and how it impacts daily living. Each question is answered on a scale of 1-5, where higher scores indicate the most impact or severity. The questionnaire responses at baseline, end of treatment and end of study will be compared.
Evaluate change in physical function from baseline through the End-of Study visit | 14 days
  * Mean change in reported physical function using the National Institute of Health (NIH) PROMIS Health Organization and PROMIS Cooperative Group questionnaire v2.0.
  * The NIH PROMIS Scale consists of 165 questions that ask the subject to rate their physical function. Each question is answered on a scale of 1-5 where higher scores indicate the lowest level of difficulty. The questionnaire responses at baseline, end of treatment and end of study will be compared.
Mean change in daily activity (step taken) from baseline | 14 days
  As measured by continuous daily wearable activity monitor
Mean change in average heart rate from baseline | 14 days
  As measured by continuous daily wearable activity monitor
Mean change in peak heart rate from baseline | 14 days
  As measured by continuous daily wearable activity monitor
Mean change in sleep duration from baseline | 14 days
  As measured by continuous daily wearable activity monitor
Mean change in sleep disturbances from baseline | 14 days
  As measured by continuous daily wearable activity monitor
Mean change in daily active minutes from baseline | 14 days
  As measured by continuous daily wearable activity monitor
Decrease in inflammatory biomarkers (CA-19 and CRP) from baseline | 6 days
  CA-19 and CRP lab results from baseline will be compared to results from Day 6
Mean change in calories consumed from baseline through the End-of-Treatment visit | 6 days
  As measured by Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool. The ASA is a system to collect 24-hour food recalls and provide complete nutrient analysis of the foods and beverages consumed during the collection timeframe. The tool is used in this study to calculate total calories consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars- Sinai Medical Center, Los Angeles, California, United States